CLINICAL TRIAL: NCT02659774
Title: Assessing the Corporate Environment in Promoting Tobacco Control and Evaluation of a Smoking Cessation Programme in Workplaces in Hong Kong
Brief Title: Smoking Cessation in Workplaces in Hong Kong [Phase II]
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Lok Sin Tong Benevolent Society, Kowloon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LSTWPLACE2015
Record Dates: First submitted 2015-07-09; First posted 2016-01-20 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Smoking
Keywords: Smoking cessation interventions
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Experimental): Health talk + workshop (Motivational intervention) + booklet + Short Message Service (SMS)
  Interventions: Behavioral: workshop (Motivational intervention); Behavioral: Health talk; Behavioral: SMS; Behavioral: Booklet
- Group B (Placebo Comparator): Face to Face counseling (Motivational intervention) + Booklet + SMS
  Interventions: Behavioral: Health talk; Behavioral: Face to Face counseling; Behavioral: SMS; Behavioral: Booklet
- Group C (Placebo Comparator): Phone counseling (Motivational intervention) + Health talk + booklet + SMS
  Interventions: Behavioral: Health talk; Behavioral: SMS; Behavioral: Booklet
- Group D (Placebo Comparator): Phone counseling (Motivational intervention) + booklet + SMS
  Interventions: Behavioral: Phone counseling; Behavioral: SMS; Behavioral: Booklet

INTERVENTIONS:
Behavioral: workshop (Motivational intervention) — Through intensive workshop which includes motivation of quitting enhancement, stress management, smoking triggers, cravings and relapse, to provide smoking cessation intervention
  Arms: Group A
Behavioral: Health talk — Health talk provided information about hazards of tobacco (active smoking, second- and third-hand smoke), benefits of quitting smoking and methods to quit smoking
  Arms: Group A; Group B; Group C
Behavioral: Face to Face counseling — Use motivational interview strategies through face-to-face counseling to provide smoking cessation intervention
  Arms: Group B
Behavioral: Phone counseling — Use motivational interview strategies through telephone counseling to provide smoking cessation intervention
  Arms: Group D
Behavioral: SMS — Use motivational interview strategies through telephone messages to provide smoking cessation intervention
Behavioral: Booklet — A 26-page booklet included information about smoking and diseases, benefits of quitting smoking, methods to quit smoking, how to handle withdrawal symptoms, stress management, declaration of quitting smoking, decisional balance of smoking or quitting

SUMMARY:
This study has the following objectives:

1. To examine the employers'/managerial staff's knowledge, attitudes and practices in promoting smoking cessation in workplace.
2. To evaluate the smoking behaviours of participants before and after attending a smoking cessation intervention.

DETAILED DESCRIPTION:
Study design In Phase I of this study, a large scale cross-sectional survey will be sent to 3000 corporations in Hong Kong. The questionnaire will examine the employers' knowledge, attitudes and practices in promoting smoking cessation in the workplace.

In Phase II, a longitudinal study will be conducted to evaluate the effectiveness of a smoking cessation intervention offered by the Department of Psychology, the University of Hong Kong. A total of 600 smokers from corporations will be recruited and interviewed before the intervention at baseline, immediately after the intervention, and at 1-, 4-, 12-, 26- and 52-week post-intervention follow-ups, in an attempt to evaluate their smoking behaviours, knowledge on smoking and satisfaction of the smoking cessation services. Self-reported quitters (did not smoke in the past 7 days) will be invited to participate in the bio-chemical validation by assessing their exhaled carbon monoxide level and the saliva cotinine level.

Process evaluation: Qualitative interviews, including in-depth interviews and/or focus group will be conducted within 1 month after 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Cantonese speaker and able to read in Chinese characters
* Smoke at least one cigarette per day
* Stay at Hong Kong during the intervention and follow-up periods (12 months)

Exclusion Criteria:

* Smokers who are psychologically or physically unable to communicate
* Smokers who are currently following other smoking cessation programme(s)
* Smokers with diagnosed psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline smoking quit rate at 6-month | 6 months after the intervention
  Quit smoking rate is defined by the self-reported 7-day point prevalence abstinence. It is a binary type (yes/no) questionnaire and participants answer the question about their smoking status in the past 7 days at 6-month after the intervention.

SECONDARY OUTCOMES:
Change from baseline smoking reduction at 6-month | 6 months after the intervention
  Smoking reduction is defined as reduced at least 50% of cigarette consumption. Participants were asked to respond to the daily cigarette consumption at 6-month after the intervention. Their daily cigarette consumption at 6-month were compared with baseline's daily cigarette consumption and determine whether they had reduced at least 50% cigarette consumption at 6-month.
Change from baseline smoking reduction at 12-month | 12 months after the intervention
  Smoking reduction is defined as reduced at least 50% of cigarette consumption. Participants were asked to respond to the daily cigarette consumption at 6-month after the intervention. Their daily cigarette consumption at 12-month were compared with baseline's daily cigarette consumption and determine whether they had reduced at least 50% cigarette consumption at 12-month.
Change from baseline smoking quit rate at 12-month | 12 months after the intervention
  Quit smoking rate is defined by the self-reported 7-day point prevalence abstinence. It is a binary type (yes/no) questionnaire and participants answer the question about their smoking status in the past 7 days at 12-month after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Man-ping Wang, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- 2/F, 61 Lung Kong Rd, Kowloon City, Lok Sin Tong Benevolent Society, Hong Kong, China